CLINICAL TRIAL: NCT02619604
Title: A Quality Improvement Approach to the Management of Chronic Lymphocytic Leukemia
Acronym: Med-IQ CLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Med-IQ (Industry); Gilead Sciences (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00063975
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-01

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinician education (Other)
  Interventions: Other: Education Intervention

INTERVENTIONS:
Other: Education Intervention — Education interventions will be delivered sporadically within the 6-month window between the time the clinician completes the pre-survey and when he/she completes the post-survey. Interventions consist of e-brief publications, teleconferences with project faculty, and evidence based resources.

SUMMARY:
This project addresses the need to improve physician knowledge and clinical practice patterns related to quality of life (QoL) concerns for patients with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
This multifaceted initiative will include evaluating patient perspectives on their QoL, evaluating provider perspectives on managing QoL, and providing education to the whole CLL care team (hematologists/oncologists, nurse practitioners, physician assistants, and nurses) on contemporary approaches for individualized, patient-centered management of CLL. Providers, including physicians, nurse practitioners, and physician assistants will participate in educational initiatives geared towards enhancing their knowledge and confidence with managing QoL concerns for patients with CLL. Pre and post surveys will be conducted with providers to evaluate change in these areas. The project aims to train this team on how to enhance communication with patients and caregivers as a means to increase patient engagement in care and QoL in this population.

ELIGIBILITY:
Inclusion Criteria: Clinician

* Participant must be a hematologist, oncologist, nurse practitioner, or physician assistant who practices medicine in the Duke Cancer Network
* Participant treats patients with CLL
* Participant is willing to participate in the educational component of this project

Inclusion Criteria: Patient

* Patient has a diagnosis of Chronic Lymphocytic Leukemia
* Patient is over the age of 18
* Patient is being treated at a Duke Cancer Network affiliate site,
* Patient is expected to see their physician or another member of their care team at least 3 times annually.
* Signed informed consent

Exclusion Criteria: Clinician

* None

Exclusion Criteria: Patient

* Patient is Non-English speaking
* Patient diagnosed with CLL < 60 days ago

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in provider knowledge with management of Quality of Life Concerns for CLL patients, as measured by survey | Baseline, 6 months
Change in provider confidence with management of Quality of Life Concerns for CLL patients, as measured by survey | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Sutton, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Network, Durham, North Carolina, United States